CLINICAL TRIAL: NCT02096601
Title: A Multicenter, Open-Label, Randomized, Dose-Finding Study Testing the Safety, Tolerability, and Pharmacokinetics (PK) of ND0612, a Liquid Formulation of Levodopa/Carbidopa (LD/CD) Delivered as a Continuous Subcutaneous Infusion (SC) in Parkinson's Disease (PD) Patients Treated With LD
Brief Title: A Safety, Tolerability, and Pharmacokinetic Study of ND0612 Delivered as a Continuous Subcutaneous in Parkinson's Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ND0612/004
Record Dates: First submitted 2014-03-18; First posted 2014-03-26 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: Motor fluctuations; levodopa pharmacokinetics; levodopa and carbidopa solution; continuous subcutaneous delivery
MeSH Terms: conditions — Parkinson Disease | interventions — entacapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ND0612L Low LD Dose (Experimental): LD daily dose equals to 115 mg administered over 8 hours SC infusion:
  * LD/CD 60/7.5 mg/mL on Study Day 3
  * LD/CD 60/14 mg/mL on Study Day 4
  * LD/CD 60/14 mg/mL and Entacapone 200 mg every 4 hours on Study Day 5
  Interventions: Drug: LD/CD SC solution; Drug: Entacapone
- ND0612H High LD Dose (Experimental): LD daily dose equals to 307 mg administered over 8 hours SC infusion:
  * LD/CD 60/7.5 mg/mL on Study Day 3
  * LD/CD 60/14 mg/mL on Study Day 4
  * LD/CD 60/14 mg/mL and Entacapone 200 mg every 4 hours on Study Day 5
  Interventions: Drug: LD/CD SC solution; Drug: Entacapone

INTERVENTIONS:
Drug: LD/CD SC solution — Levodopa/carbidopa SC solution
  Other Names: ND0612
Drug: Entacapone — Entacapone 200 mg oral tablet

SUMMARY:
An open-label randomized study to evaluate the Safety, Tolerability, and PK of Low and High single doses of ND0612 (i.e. LD/CD ratio 60/7.5 mg/mL and 60/14 mg/mL), as well as the combination with oral Entacapone (concomitant catechol-O-methyl transferase [COMT] inhibitor) in PD subjects with well-defined morning "OFF" and a good response to LD. Exploratory efficacy parameters were collected (early evidence of effectiveness as part of Phase 1).

DETAILED DESCRIPTION:
PD subjects were randomized in Low or High LD dose study group in 1:1 ratio. Each patient received singe doses ND0612 over 3 days: Day 1. LD/CD 60/7.5 mg/mL, Day 2. LD/CD 60/14 mg, and Day 3. LD/CD 60/14 mg/mL with Entacapone.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female PD patients of any race aged 30 to 80 years
2. PD diagnosis consistent with the UK PD Society Brain Bank criteria.
3. Stable doses of anti PD drugs for at least 30 days
4. PD patients with well-defined morning "OFF" and a good response to LD
5. MMSE score > 26
6. No clinically significant medical, psychiatric or laboratory abnormalities

Exclusion Criteria:

1. Atypical or secondary Parkinsonism.
2. Acute psychosis or hallucinations.
3. Subjects treated with neuroleptics
4. History of melanoma or significant skin disorders.
5. Prior neurosurgical procedure for PD.
6. Patients with a history of drug abuse or alcoholism
7. Clinically significant ECG abnormalities.
8. Renal or liver dysfunction
9. Subjects who have participated in another clinical study within 30 days

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08-11 (Actual); Primary Completion 2015-03-15 (Actual); Study Completion 2015-03-15 (Actual)

PRIMARY OUTCOMES:
Adverse events frequency | Up to 6 weeks
LD, CD and 3-OMD PK analysis from sample taken on Days 3, 4 and 5 will be used to determine the Fluctuation Index, its CV, AUC, Cmin, Cmax, and tmax. | Days 1, 2, 3 and 4
Tolerability: Number of patients who discontinued due to adverse events | Up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Medical Center, Tel Aviv